CLINICAL TRIAL: NCT00259701
Title: Transdermal Application of Acetylcholine and Nitroglycerin Without Iontophoresis.
Brief Title: Microvascular Reactivity.
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Other Study IDs: HIC-12397-1
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2005-11

CONDITIONS: Diabetes; Retinopathy; Vascular Pathology
Keywords: endothelium; iontophoresis; acetylcholine; nitroglycerin; vasodilation
MeSH Terms: conditions — Diabetes Mellitus; Retinal Diseases; Aneurysm | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: Laser Doppler Flowmetry with topical acetylcholine and nitroglycerin

SUMMARY:
This study attempts to test capillary responses to various challenges without the need for iontophoresis (electrical current).

DETAILED DESCRIPTION:
Studies of microvascular responsiveness often employ iontophoresis to fascilitate drug absorption. Iontophoresis is a confounding stimulus in such studies, and we are attempting to create tests of the microvasculature that do not require iontophoretic drug delivery.

ELIGIBILITY:
Inclusion Criteria: diabetic. -

Exclusion Criteria: not on nitrates or mydriatic eye drops within 48 hours.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: David G Silverman, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Schonberger RB, Worden WS, Shahmohammadi K, Menn K, Silverman TJ, Stout RG, Shelley KH, Silverman DG. Topical non-iontophoretic application of acetylcholine and nitroglycerin via a translucent patch: a new means for assessing microvascular reactivity. Yale J Biol Med. 2006 Mar;79(1):1-7. PMID 17876370